CLINICAL TRIAL: NCT02295800
Title: The Kabeho Study: Kigali Antiretroviral and Breastfeeding Assessment for the Elimination of HIV
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Ministry of Health, Rwanda (Other Government); University of Rwanda (Other)
Responsible Party: Sponsor
Other Study IDs: EGPAF0098
Record Dates: First submitted 2014-10-15; First posted 2014-11-20 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2014-11

CONDITIONS: Mother-to-child HIV Transmission
Keywords: HIV; PMTCT; Antenatal Care
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma specimens collected from the adult participants at the time of viral load testing and dried blood spot (DBS) specimens drawn from the infant participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mothers: HIV Infected mothers
  Interventions: Other: Standard of care; Other: Semi-structured interviews
- Infants: HIV exposed infants
  Interventions: Other: Standard of care
- Healthcare workers: Facility based healthcare workers
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Standard of care
  Groups: Infants; Mothers
Other: Semi-structured interviews
  Groups: Healthcare workers; Mothers

SUMMARY:
The study design includes an observational prospective cohort of HIV-positive pregnant/postpartum women and their infants enrolled during antenatal clinics (or immediately postpartum) from prevention of mother-to-child transmission (PMTCT) programs and followed until the infants reach the age of 18 - 24 months and semi-structure interviews with a sub-set of these women. A second study component involves semi-structured interviews with health care workers (HCW) involved in the PMTCT programs and yearly facility surveys at the selected study facilities.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Pregnant, in the last trimester of pregnancy or within two weeks post-delivery.
* Participation in the PMTCT program during antenatal care at one of the study sites
* Planning on remaining in the Kigali area after delivery
* Able and willing to give informed consent for study participation for herself and her infant(s).

If a pregnant woman is less than 18 years of age and still living with her parents, informed consent will also be required from one of her parents

Exclusion Criteria:

* Women not willing to provide informed consent to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women identified as HIV infected during antenatal care and receiving PMTCT services (regardless of ARV regimen received) in the selected antenatal clinics in Kigali, Rwanda are eligible for study enrollment. The infants born to enrolled study women during the study pregnancy will also be study participants up to the age of 18 - 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 1216 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
18 - 24 month HIV-free survival of children born to HIV-positive pregnant women | 18 - 24 months

SECONDARY OUTCOMES:
HIV-exposed infants with stunting, underweight, or wasting Infants and young children breastfed (exclusive or any breastfeeding) at various ages | 18 - 24 months
Infants and young children breastfed (exclusive or any breastfeeding) at various ages | 18 - 24 months
Adherence to the universal antiretroviral therapy (ARV) regimen among pregnant and postpartum women (Option B+) and their HIV-exposed children, including the proportion of study women with HIV RNA < 1000 copies/ml or > 2 log10 copies/mL decrease in viral | 18 - 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Emily A. Bobrow, PhD, MPH, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- Elizabeth Glaser Pediatric AIDS Foundation, Kigali, Rwanda